CLINICAL TRIAL: NCT04229303
Title: To Assess Safety, PK of Inhaled Voriconazole (ZP-059) Single Doses in Healthy Subjects (Part 1), ZP-059 Multiple Doses in Stable Asthma (Part 2) and in a Crossover Trial of ZP-059 and Oral Voriconazole Single Doses in Stable Asthma (Part 3)
Brief Title: Phase 1 Three Part SAD, MAD & Cross-Over Study of ZP-059 in Healthy and Asthmatic Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Zambon SpA (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: Z7240J01; 2019-004031-23 (EudraCT Number)
Record Dates: First submitted 2019-12-06; First posted 2020-01-18 (Actual); Results first posted 2021-11-15 (Actual); Last update posted 2021-11-15 (Actual); Status verified 2019-12

CONDITIONS: Allergic Bronchopulmonary Aspergillosis
Keywords: ABPA; Asthma; Voriconazole; Allergic Bronchopulmonary Aspergillosis
MeSH Terms: conditions — Aspergillosis, Allergic Bronchopulmonary; Asthma | interventions — Voriconazole

STUDY DESIGN:
Intervention Model Description: Safety, tolerability and PK will be assessed following either single ascending (SAD) or multiple ascending (MAD) dosing of ZP-059; Part 1 and Part 2, respectively. Part 1 will comprise 4 separate cohorts planned to receive single doses of ZP-059; part 2 will comprise 3 separate cohorts planned to receive daily doses of ZP-059 on Day 1 to 10; part 3 is a 2-period, randomised crossover study in subjects with mild to moderate stable asthma to assess the safety, tolerability and PK of single doses of ZP-059 and single doses of oral voriconazole.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (9):
- Part 1 - ZP-059 5mg (Experimental): Part 1: administration of single ascending doses (SAD) of ZP-059.
  Cohort 1: 5mg (1 x 5 mg capsule) ZP-059 single dose administered via DPI (RS01 monodose device) on Day 1.
  Interventions: Drug: Voriconazole inhaled
- Part 1 - ZP-059 10mg (Experimental): Part 1: administration of single ascending doses (SAD) of ZP-059.
  Cohort 2: 10mg (2 x 5 mg capsule) ZP-059 single dose administered via DPI (RS01 monodose device) on Day 1.
  Interventions: Drug: Voriconazole inhaled
- Part 1 - ZP-059 20mg (Experimental): Part 1: administration of single ascending doses (SAD) of ZP-059.
  Cohort 3: 20mg (4 x 5 mg capsule) ZP-059 single dose administered via DPI (RS01 monodose device) on Day 1.
  Interventions: Drug: Voriconazole inhaled
- Part 1 - ZP-059 40mg (Experimental): Part 1: administration of single ascending doses (SAD) of ZP-059.
  Cohort 4: 40mg (8 x 5 mg capsule) ZP-059 single dose administered via DPI (RS01 monodose device) on Day 1.
  Interventions: Drug: Voriconazole inhaled
- Part 2 - ZP-059 10mg bid (Experimental): Part 2: administration of multiple ascending doses (MAD) of ZP-059 on Days 1 to 10.
  Cohort 1: 10mg (2 x 5 mg capsule) ZP-059 twice daily (bid) administered via DPI (RS01 monodose device) for 9 days and once in the morning of Day 10.
  Interventions: Drug: Voriconazole inhaled
- Part 2 - ZP-059 20mg bid (Experimental): Part 2: administration of multiple ascending doses (MAD) of ZP-059 on Day 1 to 10.
  Cohort 2: 20mg (4 x 5 mg capsule) ZP-059 twice daily (bid) administered via DPI (RS01 monodose device) for 9 days and once in the morning of Day 10.
  Interventions: Drug: Voriconazole inhaled
- Part 2 - ZP-059 40mg qd (Experimental): Part 2: administration of multiple ascending doses (MAD) of ZP-059 on Day 1 to 10.
  Cohort 3: 40mg (8 x 5 mg capsule) ZP-059 once daily (qd) administered via DPI (RS01 monodose device) on Days 1 to 10.
  Interventions: Drug: Voriconazole inhaled
- Part 3 - ZP-059 / Oral Voriconazole (Experimental): Crossover treatment period: Single inhaled dose (20 mg) of ZP-059 5mg capsules administered via DPI, and a single dose of oral voriconazole (200 mg Vfend® tablet) on the morning of Day 1 of the respective treatment period with a washout period of at least 96 hours.
  Interventions: Drug: Voriconazole inhaled; Drug: oral voriconazole
- Part 3 - Oral Voriconazole / ZP-059 (Experimental): Crossover treatment period: Single dose of oral voriconazole (200 mg Vfend® tablet), and a single inhaled dose (20 mg) of ZP-059 5mg capsules administered via DPI on the morning of Day 1 of the respective treatment period with a washout period of at least 96 hours.
  Interventions: Drug: Voriconazole inhaled; Drug: oral voriconazole

INTERVENTIONS:
Drug: Voriconazole inhaled — Part 1 (SAD): eligible subjects received a single ascending inhaled dose (5 mg, 10 mg, 20 mg, and 40 mg) of ZP-059 5mg capsules administered via dry powder inhaler (DPI) on the morning of Day 1.
  Part 2 (MAD): eligible subjects received 2 (10mg twice daily [BID]) or 4 [20mg BID]) inhaled doses of ZP-059 5mg capsules administered via DPI BID for 9 days and once in the morning of Day 10, or 8 inhaled doses of ZP-059 5 mg capsules (40mg once daily [QD]) for 10 days. For QD dosing, subjects received QD doses of ZP-059 (at hour 0) on Days 1 to 10.
  Part 3 (2-period crossover): eligible subjects received a 4 [20mg BID] inhaled doses of ZP-059 5mg capsules administered via DPI on the morning of Day 1 according to the crossover scheme of the study.
  ZP-059 (inhaled voriconazole) was provided in clear, colorless size 3 hydroxypropylmethylcellulose hard capsules, which were individually and manually triggered by a breath actuated inhalation device (RS01 monodose inhaler).
  Other Names: ZP-059
Drug: oral voriconazole — Part 3 (2-period crossover): eligible subjects received a single dose of oral voriconazole (200mg oral film-coated tablet, Vfend) on the morning of Day 1 according to the crossover scheme of the study.
  Other Names: Vfend
  Arms: Part 3 - Oral Voriconazole / ZP-059; Part 3 - ZP-059 / Oral Voriconazole

SUMMARY:
The primary safety objectives were:

* Part 1: To determine the safety and tolerability of single doses of ZP-059 in healthy subjects
* Part 2: To determine the safety and tolerability of multiple doses of ZP-059 in subjects with mild stable asthma
* Part 3: To determine the safety and tolerability of single doses of ZP-059 in subjects with mild to moderate stable asthma.

The primary PK objectives were:

* Part 1: To characterize systemic PK of voriconazole and N-oxide voriconazole after single doses of ZP-059 in healthy subjects
* Part 2: To characterize systemic PK of voriconazole and N-oxide voriconazole after multiple doses of ZP-059 in subjects with mild stable asthma
* Part 3: To characterize systemic PK of voriconazole and N-oxide voriconazole after single doses of ZP-059 and single doses of oral voriconazole in subjects with mild to moderate stable asthma.

DETAILED DESCRIPTION:
This was an integrated Phase 1, single centre, multi-part, open-label study in both healthy subjects (Part 1), subjects with mild stable asthma (Part 2) and subjects with mild to moderate stable asthma (Part 3). In all three parts of the study every effort was made to include as close as possible an equal balance between male and female subjects.

This study assessed safety, tolerability and PK of single and multiple ascending doses of ZP-059 capsules administered as dry powder for inhalation in Part 1 to healthy volunteers (single ascending dose; SAD) and in Part 2 to subjects with mild asthma (multiple ascending dose; MAD), respectively.

In Part 3, the bioavailability of ZP-059 in subjects with mild to moderate stable asthma were compared to that of oral voriconazole. Part 3 started only after review of safety data from cohorts 1 to 4 of Part 1 (SAD) have been completed. Parts 2 and 3 of the study also explored voriconazole concentrations in induced sputum samples in asthmatic subjects.

As part of the safety and tolerability assessment, this study investigated the effects of ZP-059 on airway function in both mild and mild to moderate stable asthma subjects.

ELIGIBILITY:
Inclusion Criteria (part 1):

* Female subjects must be either of non-childbearing potential or if of childbearing potential use a highly effective birth control method
* Male subjects with female partners of childbearing potential must be vasectomised with documented medical assessment of the surgical success or use highly effective contraception together with their female partner(s)
* Subject must agree not to donate semen or ova/oocytes during the study and for 14 days after the last dose of IMP.
* BMI ≥ 18.0 and ≤ 35.0 kg/m2 at Screening.
* Are willing and able to comply with all aspects of the protocol.
* FEV1 ≥80% of the predicted value and FEV1/FVC ratio > 0.70; at screening.
* Able to demonstrate the correct inhalation technique for use of delivery device during the study at screening and pre-dose Day 1.

Inclusion Criteria (part 2):

* Subjects with mild stable asthma with a documented physician confirmed diagnosis of asthma for at least 3 months prior to screening.
* Asthma assessed by investigator as being stable for at least 4 weeks prior to screening and prior to Day 1.
* Female subjects must be either of non-childbearing potential or if of childbearing potential use a highly effective birth control method
* Male subjects with female partners of childbearing potential must be vasectomised with documented medical assessment of the surgical success or use highly effective contraception together with their female partner(s).
* Subject must agree not to donate semen or ova/oocytes during the study and for 14 days after the last dose of IMP.
* Body mass index (BMI) ≥ 18.0 and ≤ 35.0 kg/m2 at Screening.
* Are willing and able to comply with all aspects of the protocol.
* Subject is being treated with short acting beta-agonists alone or in conjunction with low to medium doses of ICS.
* Pre-bronchodilator FEV1 ≥70% of the predicted value at screening.
* Able to demonstrate the correct inhalation technique for use of delivery device during the study at screening and pre-dose Day 1.

Inclusion Criteria (part 3):

* Subjects with mild to moderate stable asthma with a documented physician confirmed diagnosis of asthma for at least 3 months prior to screening.
* Asthma assessed by investigator as being stable for at least 4 weeks prior to screening and prior to randomisation.
* Female subjects must be either of non-childbearing potential or if of childbearing potential use a highly effective birth control method .
* Male subjects with female partners of childbearing potential must be vasectomised with documented medical assessment of the surgical success or use highly effective contraception together with their female partner(s)
* Subject must agree not to donate semen or ova/oocytes during the study and for 14 days after the last dose of IMP.
* BMI ≥ 18.0 and ≤ 35.0 kg/m2 at Screening.
* Are willing and able to comply with all aspects of the protocol.
* Subject is being treated with low to medium doses of ICS with or without long-acting beta-agonists.
* Pre-bronchodilator FEV1 ≥70% of the predicted value at screening.
* Able to demonstrate the correct inhalation technique for use of delivery device during the study at screening and pre-dose Day 1, Treatment Period 1.
* Able to produce a sputum sample with a minimum weight of 50 mg at screening.

Exclusion Criteria (part 1):

* Subjects who are Chinese or Japanese.
* Subjects who have received any IMP in a clinical research study within the previous 3 months prior to Day 1.
* Participation in other interventional studies for the duration of the study.
* Subjects who are study site employees or immediate family members of a study site or sponsor employee.
* History of any drug or alcohol abuse in the past 2 years prior to screening.
* Regular alcohol consumption in males >21 units per week and females >14 units per week (1 unit = ½ pint beer, a 25 mL shot of 40% spirit or a 125 mL glass of wine depending on type).
* Current tobacco or marijuana smokers and those who have smoked within the last 12 months prior to screening or prior to Day 1.
* A confirmed positive urine cotinine test at screening or Day -1.
* Current users of e-cigarettes or nicotine replacement products and those who have used these products within the last 12 months prior to screening or prior to Day 1.
* Smoking history of >5 pack years at screening.
* Females of childbearing potential who are pregnant or lactating, or who plan to become pregnant during the study. A woman is considered of childbearing potential unless she is permanently sterile (hysterectomy, bilateral salpingectomy, bilateral oophorectomy, bilateral tubal occlusion/ligation) or is postmenopausal (had no menses for 12 months without an alternative medical cause).
* Female subject with a positive pregnancy test at screening or pre-dose on Day 1.
* Subjects who do not have suitable veins for multiple venepunctures/cannulation as assessed by the investigator at screening.
* Evidence or history of clinically significant abnormal biochemistry, haematology or urinalysis at screening, as judged by the investigator; the investigator should contact the medical monitor and /or the sponsor if required.
* Positive urine drugs of abuse test or alcohol breath test result at screening or Day -1.
* History of or currently infected with/carrier of human immunodeficiency virus (HIV).
* Positive hepatitis B surface antigen (HBsAg), hepatitis C virus antibody (HCV Ab) or human immunodeficiency virus (HIV) results. Subjects who are HBs antibody positive or HB core antibody positive are not excluded provided the HBsAg result is negative. Subjects who are HCV Ab positive are not excluded if a subsequent HCV RNA test is negative.
* Evidence or history of clinically significant cardiovascular, renal, hepatic, endocrine, immunological or autoimmune, dermatological, ophthalmological, chronic respiratory or gastrointestinal disease, neurological or psychiatric disorder, as judged by the investigator.
* Subjects with congestive heart failure or a history of congestive heart failure.
* 12-lead ECGs demonstrating a mean QTcF interval >450 msec for males or QTcF interval >470 msec for females at screening or pre-dose Day 1.
* History of severe cough or bronchospasm upon inhalation of any inhalation product.
* Serious adverse reaction or serious hypersensitivity to any drug or the formulation excipients.
* Have had allergies to or hypersensitivity reactions after administration of voriconazole or other antifungal azoles.
* Presence or history of clinically significant allergy, including drug allergies, but excluding untreated, mild seasonal allergies, as judged by the investigator. Hay fever is allowed unless it is active.
* Major trauma or surgery within the last 3 months prior to screening or prior to Day 1.
* Planned or elective surgery or hospitalisations for the duration of the study that may interfere with study logistics or safety.
* Donation or loss of more than 400 mL of blood within the previous 3 months prior to screening.
* Subjects who are taking, or have taken, any prescribed or over-the-counter drug (other than ≤4 g per day of paracetamol, hormonal contraception or hormone replacement therapy), dietary supplements or CYP3A4 or CYP2C19 inhibitors in the 14 days (or 5 half-lives, whichever is longer) prior to Day 1 and for the duration of the study. Exceptions may apply on a case by case basis, if considered not to interfere with the objectives of the study, as agreed by the Principal Investigator and sponsor's medical monitor.
* Subjects who are taking or have taken any herbal remedies or CYP3A4 or CYP2C19 inducers in the 28 days prior to Day 1.
* Any use of voriconazole in the 3 months prior to Day 1.
* Subjects who have received a live or killed/inactive vaccine in the 14 days prior to Day 1.
* Upper respiratory tract infection (excluding otitis media), fever, acute or chronic cough within 14 days of Day 1, or lower respiratory tract infection within the last 4 weeks prior to Day 1.
* Recent (within the last 4 weeks prior to Day 1) clinically significant bacterial, viral or fungal infection that required systemic (oral or intravenous) antibiotics, antivirals or antifungals; topical treatments, other than antifungals, are allowed.
* Other social, psychiatric, surgical or medical conditions, or screening laboratory abnormalities that may increase subject risk associated with study participation or may interfere with the interpretation of study results and, in the judgement of the investigator would make the subject inappropriate for entry into the study.
* Failure to satisfy the investigator of fitness to participate for any reason.

Exclusion Criteria (part 2 and 3):

* Subjects who are Chinese or Japanese.
* Subjects who have received any IMP in a clinical research study within the previous 3 months prior to Day 1.
* Participation in other interventional studies for the duration of the study.
* Subjects who are study site employees, or immediate family members of a study site or sponsor employee.
* Subjects who have previously received IMP in this study.
* History of any drug or alcohol abuse in the past 2 years prior to screening.
* Regular alcohol consumption in males >21 units per week and females >14 units per week (1 unit = ½ pint beer, a 25 mL shot of 40% spirit or a 125 mL glass of wine depending on type).
* Current tobacco or marijuana smokers and those who have smoked within the last 12 months prior to screening or prior to Day 1.
* A confirmed positive urine cotinine test at screening or Day -1.
* Current users of e-cigarettes or nicotine replacement products and those who have used these products within the last 12 months prior to screening or prior to Day 1.
* Smoking history of >5 pack years at screening.
* Females of childbearing potential who are pregnant or lactating, or who plan to become pregnant during the study. A woman is considered of childbearing potential unless she is permanently sterile (hysterectomy, bilateral salpingectomy, bilateral oophorectomy, bilateral tubal occlusion/ligation) or is postmenopausal (had no menses for 12 months without an alternative medical cause).
* Female subject with a positive pregnancy test at screening or pre-dose Day 1.
* Subjects who do not have suitable veins for multiple venepunctures/cannulation as assessed by the investigator at screening.
* Evidence or history of clinically significant abnormal biochemistry, haematology or urinalysis at screening, as judged by the investigator; the investigator should contact the medical monitor and /or the sponsor if required.
* Positive urine drugs of abuse test result (unless in the opinion of the investigator this can be explained by the subject's current medications) at screening or Day -1; unexpected positive results may require discussion with sponsor).
* Positive alcohol breath test at screening or Day -1.
* History of or currently infected with/carrier of HIV.
* Positive HBsAg, HCV Ab or HIV results. Subjects who are HBs antibody positive or HB core antibody positive are not excluded provided the HBsAg result is negative. Subjects who are HCV Ab positive are not excluded if a subsequent HCV RNA test is negative.
* Evidence or history of clinically significant cardiovascular, renal, hepatic, dermatologic, ophthalmologic or gastrointestinal disease, neurological or psychiatric disorder, as judged by the investigator.
* Evidence of history of endocrine, immunological, autoimmune disease that would affect the subject's safety or confound the assessment of study endpoints in the opinion of the investigator.
* Current diagnosis of any chronic airways disease other than asthma such as Chronic Obstructive Pulmonary Disease, pulmonary fibrosis, CF, Churg-Strauss syndrome, bronchiectasis.
* Evidence of ventricular dysfunction such as congestive cardiac failure (CCF) or a history of CCF assessed at screening and pre-dose Day 1.
* 12-lead ECG demonstrating a mean QTcF interval >450 msec for males or >470 msec for females at screening or pre-dose Day 1.
* Serious adverse reaction or serious hypersensitivity to any drug or the formulation excipients.
* Have had allergies to or hypersensitivity reactions after administration of voriconazole or other antifungal azoles.
* Presence or history of clinically significant allergy, including drug allergies, as judged by the investigator. Hay fever is allowed unless it is active.
* Major trauma or surgery within the last 3 months prior to screening or prior to Day 1.
* Planned or elective surgery, hospitalisations for the duration of the study that may interfere with study logistics or safety.
* Donation or loss of more than 400 mL of blood within the previous 3 months prior to screening.
* Subjects who are taking, or have taken, any prescribed or over-the-counter drugs that are CYP3A4 or CYP2C19 inhibitors in the 14 days (or 5 half-lives, whichever is longer) prior to Day 1 and for the duration of the study.
* Subjects who are taking or have taken any herbal remedies or CYP3A4 or CYP2C19 inducers in the 28 days prior to Day 1.
* Subjects who have received a live or killed/inactive vaccine in the 14 days prior to Day 1.
* Presence of hoarseness or oropharyngeal candidiasis at screening or prior to dosing on Day 1.
* Any use of voriconazole in the 3 months prior to Day 1.
* History of life-threatening asthma, defined as an asthma episode that required intubation and/or was associated with hypercapnia, respiratory arrest and/or hypoxic seizures.
* Hospitalisation (including accident and emergency visits) for the treatment of asthma within 3 months prior to screening or prior to Day 1 or have been hospitalised or have attended the accident and emergency for asthma more than twice in the 12 months prior to screening.
* Occurrence of asthma exacerbations or respiratory tract infections within 4 weeks prior to screening or prior to Day 1.
* Recent (within the last 4 weeks prior to Day 1) clinically significant bacterial, viral or fungal infection that required systemic (oral or intravenous) antibiotics, antivirals or antifungals; topical treatments, other than antifungals, are allowed.
* Other social, psychiatric, surgical or medical conditions, or screening laboratory abnormalities that may increase subject risk associated with study participation or may interfere with the interpretation of study results and, in the judgement of the Investigator would make the subject inappropriate for entry into the study.
* Failure to satisfy the investigator of fitness to participate for any reason.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 58 (Actual)
Dates: Start 2020-02-11 (Actual); Primary Completion 2020-08-31 (Actual); Study Completion 2020-08-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sukh Dave Singh, Prof, MD,, Study Director — The Medicine Evaluation Unit (MEU) Ltd, Langley building,
Locations (1):
- Medicines Evaluation Unit Ltd. (MEU), Manchester, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Caponetti G, Sala F, Cervetti A, Colombo D, Tiberio E, Singh D. Phase I Study of the Safety, Tolerability, and Pharmacokinetics of Inhaled Voriconazole in Healthy Volunteers and Subjects With Stable Asthma. Pharmacol Res Perspect. 2025 Feb;13(1):e70064. doi: 10.1002/prp2.70064. PMID 39918069

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The investigator or his/her representative explained the nature of the study to the subject and answered all questions regarding the study. Subjects had to be informed that their participation was voluntary. Subjects were required to sign a statement of informed consent that met the requirements of UK regulations, ICH E6 GCP guidelines, General Data Protection Regulation, and the IEC or study site requirements.
  The authorized person who obtained the informed consent had to also sign the ICF.
Pre-assignment Details: Subjects were screened for eligibility to participate in the study within 28 days before dosing (Day 1). Part 2 and Part 3 subjects who had completed the initial screening visit attended the study site on Day -4 or Day -3, for Covid-19 reverse transcriptase - polymerase chain reaction (RT-PCR) test, together with additional daily tympanic temperature measurements, and other tests as applicable.
  Subjects were then be admitted to the study site on the evening of Day -1.
Groups:
- Part 1 - ZP-059 5mg: Part 1: administration of single ascending doses (SAD) of ZP-059.
  Cohort 1: 5mg (1 x 5 mg capsule) ZP-059 single dose administered via DPI (RS01 monodose device) on Day 1.
  Voriconazole inhaled: Part 1 (SAD): eligible subjects received a single ascending inhaled dose (5 mg, 10 mg, 20 mg, and 40 mg) of ZP-059 5mg capsules administered via dry powder inhaler (DPI) on the morning of Day 1.
  Part 2 (MAD): eligible subjects received 2 (10mg twice daily [BID]) or 4 [20mg BID]) inhaled doses of ZP-059 5mg capsules administered via DPI BID for 9 days and once in the morning of Day 10, or 8 inhaled doses of ZP-059 5 mg capsules (40mg once daily [QD]) for 10 days. For QD dosing, subjects received QD doses of ZP-059 (at hour 0) on Days 1 to 10.
  Part 3 (2-period crossover): eligible subjects received a single inhaled dose (20mg) of ZP-059 5mg capsules administered via DPI on the morning of Day 1 according to the crossover scheme of the study.
  ZP-059 (inhaled voriconazole) was provided in clear, colorless size 3 hydroxypropylmethylcellulose hard capsules, which were individually and manually triggered by a breath actuated inhalation device (RS01 monodose inhaler).
- Part 1 - ZP-059 10mg: Part 1: administration of single ascending doses (SAD) of ZP-059.
  Cohort 2: 10mg (2 x 5 mg capsule) ZP-059 single dose administered via DPI (RS01 monodose device) on Day 1.
  Voriconazole inhaled: Part 1 (SAD): eligible subjects received a single ascending inhaled dose (5 mg, 10 mg, 20 mg, and 40 mg) of ZP-059 5mg capsules administered via dry powder inhaler (DPI) on the morning of Day 1.
  Part 2 (MAD): eligible subjects received 2 (10mg twice daily [BID]) or 4 [20mg BID]) inhaled doses of ZP-059 5mg capsules administered via DPI BID for 9 days and once in the morning of Day 10, or 8 inhaled doses of ZP-059 5 mg capsules (40mg once daily [QD]) for 10 days. For QD dosing, subjects received QD doses of ZP-059 (at hour 0) on Days 1 to 10.
  Part 3 (2-period crossover): eligible subjects received a single inhaled dose (20mg) of ZP-059 5mg capsules administered via DPI on the morning of Day 1 according to the crossover scheme of the study.
  ZP-059 (inhaled voriconazole) was provided in clear, colorless size 3 hydroxypropylmethylcellulose hard capsules, which were individually and manually triggered by a breath actuated inhalation device (RS01 monodose inhaler).
- Part 1 - ZP-059 20mg: Part 1: administration of single ascending doses (SAD) of ZP-059.
  Cohort 3: 20mg (4 x 5 mg capsule) ZP-059 single dose administered via DPI (RS01 monodose device) on Day 1.
  Voriconazole inhaled: Part 1 (SAD): eligible subjects received a single ascending inhaled dose (5 mg, 10 mg, 20 mg, and 40 mg) of ZP-059 5mg capsules administered via dry powder inhaler (DPI) on the morning of Day 1.
  Part 2 (MAD): eligible subjects received 2 (10mg twice daily [BID]) or 4 [20mg BID]) inhaled doses of ZP-059 5mg capsules administered via DPI BID for 9 days and once in the morning of Day 10, or 8 inhaled doses of ZP-059 5 mg capsules (40mg once daily [QD]) for 10 days. For QD dosing, subjects received QD doses of ZP-059 (at hour 0) on Days 1 to 10.
  Part 3 (2-period crossover): eligible subjects received a single inhaled dose (20mg) of ZP-059 5mg capsules administered via DPI on the morning of Day 1 according to the crossover scheme of the study.
  ZP-059 (inhaled voriconazole) was provided in clear, colorless size 3 hydroxypropylmethylcellulose hard capsules, which were individually and manually triggered by a breath actuated inhalation device (RS01 monodose inhaler).
- Part 1 - ZP-059 40mg: Part 1: administration of single ascending doses (SAD) of ZP-059.
  Cohort 4: 40mg (8 x 5 mg capsule) ZP-059 single dose administered via DPI (RS01 monodose device) on Day 1.
  Voriconazole inhaled: Part 1 (SAD): eligible subjects received a single ascending inhaled dose (5 mg, 10 mg, 20 mg, and 40 mg) of ZP-059 5mg capsules administered via dry powder inhaler (DPI) on the morning of Day 1.
  Part 2 (MAD): eligible subjects received 2 (10mg twice daily [BID]) or 4 [20mg BID]) inhaled doses of ZP-059 5mg capsules administered via DPI BID for 9 days and once in the morning of Day 10, or 8 inhaled doses of ZP-059 5 mg capsules (40mg once daily [QD]) for 10 days. For QD dosing, subjects received QD doses of ZP-059 (at hour 0) on Days 1 to 10.
  Part 3 (2-period crossover): eligible subjects received a single inhaled dose (20mg) of ZP-059 5mg capsules administered via DPI on the morning of Day 1 according to the crossover scheme of the study.
  ZP-059 (inhaled voriconazole) was provided in clear, colorless size 3 hydroxypropylmethylcellulose hard capsules, which were individually and manually triggered by a breath actuated inhalation device (RS01 monodose inhaler).
- Part 2 - ZP-059 10mg Bid: Part 2: administration of multiple ascending doses (MAD) of ZP-059 on Days 1 to 10.
  Cohort 1: 10mg (2 x 5 mg capsule) ZP-059 twice daily (bid) administered via DPI (RS01 monodose device) for 9 days and once in the morning of Day 10.
  Voriconazole inhaled: Part 1 (SAD): eligible subjects received a single ascending inhaled dose (5 mg, 10 mg, 20 mg, and 40 mg) of ZP-059 5mg capsules administered via dry powder inhaler (DPI) on the morning of Day 1.
  Part 2 (MAD): eligible subjects received 2 (10mg twice daily [BID]) or 4 [20mg BID]) inhaled doses of ZP-059 5mg capsules administered via DPI BID for 9 days and once in the morning of Day 10, or 8 inhaled doses of ZP-059 5 mg capsules (40mg once daily [QD]) for 10 days. For QD dosing, subjects received QD doses of ZP-059 (at hour 0) on Days 1 to 10.
  Part 3 (2-period crossover): eligible subjects received a single inhaled dose (20mg) of ZP-059 5mg capsules administered via DPI on the morning of Day 1 according to the crossover scheme of the study.
  ZP-059 (inhaled voriconazole) was provided in clear, colorless size 3 hydroxypropylmethylcellulose hard capsules, which were individually and manually triggered by a breath actuated inhalation device (RS01 monodose inhaler).
- Part 2 - ZP-059 20mg Bid: Part 2: administration of multiple ascending doses (MAD) of ZP-059 on Day 1 to 10.
  Cohort 2: 20mg (4 x 5 mg capsule) ZP-059 twice daily (bid) administered via DPI (RS01 monodose device) for 9 days and once in the morning of Day 10.
  Voriconazole inhaled: Part 1 (SAD): eligible subjects received a single ascending inhaled dose (5 mg, 10 mg, 20 mg, and 40 mg) of ZP-059 5mg capsules administered via dry powder inhaler (DPI) on the morning of Day 1.
  Part 2 (MAD): eligible subjects received 2 (10mg twice daily [BID]) or 4 [20mg BID]) inhaled doses of ZP-059 5mg capsules administered via DPI BID for 9 days and once in the morning of Day 10, or 8 inhaled doses of ZP-059 5 mg capsules (40mg once daily [QD]) for 10 days. For QD dosing, subjects received QD doses of ZP-059 (at hour 0) on Days 1 to 10.
  Part 3 (2-period crossover): eligible subjects received a single inhaled dose (20mg) of ZP-059 5mg capsules administered via DPI on the morning of Day 1 according to the crossover scheme of the study.
  ZP-059 (inhaled voriconazole) was provided in clear, colorless size 3 hydroxypropylmethylcellulose hard capsules, which were individually and manually triggered by a breath actuated inhalation device (RS01 monodose inhaler).
- Part 2 - ZP-059 40mg qd: Part 2: administration of multiple ascending doses (MAD) of ZP-059 on Day 1 to 10.
  Cohort 3: 40mg (8 x 5 mg capsule) ZP-059 once daily (qd) d) administered via DPI (RS01 monodose device) on Days 1 to 10.
  Voriconazole inhaled: Part 1 (SAD): eligible subjects received a single ascending inhaled dose (5 mg, 10 mg, 20 mg, and 40 mg) of ZP-059 5mg capsules administered via dry powder inhaler (DPI) on the morning of Day 1.
  Part 2 (MAD): eligible subjects received 2 (10mg twice daily [BID]) or 4 [20mg BID]) inhaled doses of ZP-059 5mg capsules administered via DPI BID for 9 days and once in the morning of Day 10, or 8 inhaled doses of ZP-059 5 mg capsules (40mg once daily [QD]) for 10 days. For QD dosing, subjects received QD doses of ZP-059 (at hour 0) on Days 1 to 10.
  Part 3 (2-period crossover): eligible subjects received a single inhaled dose (20mg) of ZP-059 5mg capsules administered via DPI on the morning of Day 1 according to the crossover scheme of the study.
  ZP-059 (inhaled voriconazole) was provided in clear, colorless size 3 hydroxypropylmethylcellulose hard capsules, which were individually and manually triggered by a breath actuated inhalation device (RS01 monodose inhaler).
- Part 3 - ZP-059 / Oral Voriconazole: Crossover treatment period: Single inhaled dose (20 mg) of ZP-059 5mg capsules administered via DPI, and a single dose of oral voriconazole (200 mg Vfend® tablet) on the morning of Day 1 of the respective treatment period with a washout period of at least 96 hours.
  Voriconazole inhaled: Part 1 (SAD): eligible subjects received a single ascending inhaled dose (5 mg, 10 mg, 20 mg, and 40 mg) of ZP-059 5mg capsules administered via dry powder inhaler (DPI) on the morning of Day 1.
  Part 2 (MAD): eligible subjects received 2 (10mg twice daily [BID]) or 4 [20mg BID]) inhaled doses of ZP-059 5mg capsules administered via DPI BID for 9 days and once in the morning of Day 10, or 8 inhaled doses of ZP-059 5 mg capsules (40mg once daily [QD]) for 10 days. For QD dosing, subjects received QD doses of ZP-059 (at hour 0) on Days 1 to 10.
  Part 3 (2-period crossover): eligible subjects received a single inhaled dose (20mg) of ZP-059 5mg capsules administered via DPI on the morning of Day 1 according to the crossover scheme of the study.
  ZP-059 (inhaled voriconazole) was provided in clear, colorless size 3 hydroxypropylmethylcellulose hard capsules, which were individually and manually triggered by a breath actuated inhalation device (RS01 monodose inhaler).
  oral voriconazole: Part 3 (2-period crossover): eligible subjects received a single dose of oral voriconazole (200mg oral film-coated tablet, Vfend) on the morning of Day 1 according to the crossover scheme of the study.
- Part 3 - Oral Voriconazole / ZP-059: Crossover treatment period: Single dose of oral voriconazole (200 mg Vfend® tablet), and a single inhaled dose (20 mg) of ZP-059 5mg capsules administered via DPI on the morning of Day 1 of the respective treatment period with a washout period of at least 96 hours.
  Voriconazole inhaled: Part 1 (SAD): eligible subjects received a single ascending inhaled dose (5 mg, 10 mg, 20 mg, and 40 mg) of ZP-059 5mg capsules administered via dry powder inhaler (DPI) on the morning of Day 1.
  Part 2 (MAD): eligible subjects received 2 (10mg twice daily [BID]) or 4 [20mg BID]) inhaled doses of ZP-059 5mg capsules administered via DPI BID for 9 days and once in the morning of Day 10, or 8 inhaled doses of ZP-059 5 mg capsules (40mg once daily [QD]) for 10 days. For QD dosing, subjects received QD doses of ZP-059 (at hour 0) on Days 1 to 10.
  Part 3 (2-period crossover): eligible subjects received a single inhaled dose (20mg) of ZP-059 5mg capsules administered via DPI on the morning of Day 1 according to the crossover scheme of the study.
  ZP-059 (inhaled voriconazole) was provided in clear, colorless size 3 hydroxypropylmethylcellulose hard capsules, which were individually and manually triggered by a breath actuated inhalation device (RS01 monodose inhaler).
  oral voriconazole: Part 3 (2-period crossover): eligible subjects received a single dose of oral voriconazole (200mg oral film-coated tablet, Vfend) on the morning of Day 1 according to the crossover scheme of the study.
Period: Overall Study
Arm/Group | Part 1 - ZP-059 5mg | Part 1 - ZP-059 10mg | Part 1 - ZP-059 20mg | Part 1 - ZP-059 40mg | Part 2 - ZP-059 10mg Bid | Part 2 - ZP-059 20mg Bid | Part 2 - ZP-059 40mg qd | Part 3 - ZP-059 / Oral Voriconazole | Part 3 - Oral Voriconazole / ZP-059
Started | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 8 | 8
Completed | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 8 | 8
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Enrolled Set: subjects who passed screening irrespective of whether they received study treatment.
Groups:
- Part 2 - ZP-059 40mg qd: Part 2: administration of multiple ascending doses (MAD) of ZP-059 on Day 1 to 10.
  Cohort 3: 40mg (8 x 5 mg capsule) ZP-059 once daily (qd) administered via DPI (RS01 monodose device) on Days 1 to 10.
  Voriconazole inhaled: Part 1 (SAD): eligible subjects received a single ascending inhaled dose (5 mg, 10 mg, 20 mg, and 40 mg) of ZP-059 5mg capsules administered via dry powder inhaler (DPI) on the morning of Day 1.
  Part 2 (MAD): eligible subjects received 2 (10mg twice daily [BID]) or 4 [20mg BID]) inhaled doses of ZP-059 5mg capsules administered via DPI BID for 9 days and once in the morning of Day 10, or 8 inhaled doses of ZP-059 5 mg capsules (40mg once daily [QD]) for 10 days. For QD dosing, subjects received QD doses of ZP-059 (at hour 0) on Days 1 to 10.
  Part 3 (2-period crossover): eligible subjects received a single inhaled dose (20mg) of ZP-059 5mg capsules administered via DPI on the morning of Day 1 according to the crossover scheme of the study.
  ZP-059 (inhaled voriconazole) was provided in clear, colorless size 3 hydroxypropylmethylcellulose hard capsules, which were individually and manually triggered by a breath actuated inhalation device (RS01 monodose inhaler).
- Total: Total of all reporting groups
Arm/Group | Part 1 - ZP-059 5mg | Part 1 - ZP-059 10mg | Part 1 - ZP-059 20mg | Part 1 - ZP-059 40mg | Part 2 - ZP-059 10mg Bid | Part 2 - ZP-059 20mg Bid | Part 2 - ZP-059 40mg qd | Part 3 - ZP-059 / Oral Voriconazole | Part 3 - Oral Voriconazole / ZP-059 | Total
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 8 | 8 | 58
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 8 | 8 | 58
  >=65 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 3 | 3 | 2 | 2 | 2 | 3 | 1 | 2 | 21
  Male | 3 | 3 | 3 | 4 | 4 | 4 | 3 | 7 | 6 | 37
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 2
  White | 6 | 5 | 6 | 6 | 5 | 5 | 6 | 6 | 7 | 52
  More than one race | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United Kingdom | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 8 | 8 | 58

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-Emergent Adverse Events (TEAE)
Description: An AE is any untoward medical occurrence in a patient or clinical study subject, temporally associated with the use of IMP, whether or not considered related to the study IMP.
Time Frame: Part 1: screening (Day -28 to -1) to follow-up (8 to 12 days after last dose); part 2: screening (Day -28 to -1) to follow-up (11-17 days after last dose); Part 3: screening (Day -28 to -1) to follow-up (8-12 days after last dose of study drug).
Population: Safety Analysis Set (SAF): subjects who received at least 1 IMP dose, analyzed according to the treatment actually taken.
Measure: Number; unit: participants
Groups:
- Part 3 - ZP-059 20mg: Crossover treatment period: Single inhaled dose (20 mg) of ZP-059 5mg capsules administered via DPI, and a single dose of oral voriconazole (200 mg Vfend® tablet) on the morning of Day 1 of the respective treatment period with a washout period of at least 96 hours.
  Voriconazole inhaled: Part 1 (SAD): eligible subjects received a single ascending inhaled dose (5 mg, 10 mg, 20 mg, and 40 mg) of ZP-059 5mg capsules administered via dry powder inhaler (DPI) on the morning of Day 1.
  Part 2 (MAD): eligible subjects received 2 (10mg twice daily [BID]) or 4 [20mg BID]) inhaled doses of ZP-059 5mg capsules administered via DPI BID for 9 days and once in the morning of Day 10, or 8 inhaled doses of ZP-059 5 mg capsules (40mg once daily [QD]) for 10 days. For QD dosing, subjects received QD doses of ZP-059 (at hour 0) on Days 1 to 10.
  Part 3 (2-period crossover): eligible subjects received a single inhaled dose (20mg) of ZP-059 5mg capsules administered via DPI on the morning of Day 1 according to the crossover scheme of the study.
  ZP-059 (inhaled voriconazole) was provided in clear, colorless size 3 hydroxypropylmethylcellulose hard capsules, which were individually and manually triggered by a breath actuated inhalation device (RS01 monodose inhaler).
  oral voriconazole: Part 3 (2-period crossover): eligible subjects received a single dose of oral voriconazole (200mg oral film-coated tablet, Vfend) on the morning of Day 1 according to the crossover scheme of the study.
- Part 3 - Oral Voriconazole 200mg: Crossover treatment period: Single dose of oral voriconazole (200 mg Vfend® tablet), and a single inhaled dose (20 mg) of ZP-059 5mg capsules administered via DPI on the morning of Day 1 of the respective treatment period with a washout period of at least 96 hours.
  Voriconazole inhaled: Part 1 (SAD): eligible subjects received a single ascending inhaled dose (5 mg, 10 mg, 20 mg, and 40 mg) of ZP-059 5mg capsules administered via dry powder inhaler (DPI) on the morning of Day 1.
  Part 2 (MAD): eligible subjects received 2 (10mg twice daily [BID]) or 4 [20mg BID]) inhaled doses of ZP-059 5mg capsules administered via DPI BID for 9 days and once in the morning of Day 10, or 8 inhaled doses of ZP-059 5 mg capsules (40mg once daily [QD]) for 10 days. For QD dosing, subjects received QD doses of ZP-059 (at hour 0) on Days 1 to 10.
  Part 3 (2-period crossover): eligible subjects received a single inhaled dose (20mg) of ZP-059 5mg capsules administered via DPI on the morning of Day 1 according to the crossover scheme of the study.
  ZP-059 (inhaled voriconazole) was provided in clear, colorless size 3 hydroxypropylmethylcellulose hard capsules, which were individually and manually triggered by a breath actuated inhalation device (RS01 monodose inhaler).
  oral voriconazole: Part 3 (2-period crossover): eligible subjects received a single dose of oral voriconazole (200mg oral film-coated tablet, Vfend) on the morning of Day 1 according to the crossover scheme of the study.
Arm/Group | Part 1 - ZP-059 5mg | Part 1 - ZP-059 10mg | Part 1 - ZP-059 20mg | Part 1 - ZP-059 40mg | Part 2 - ZP-059 10mg Bid | Part 2 - ZP-059 20mg Bid | Part 2 - ZP-059 40mg qd | Part 3 - ZP-059 20mg | Part 3 - Oral Voriconazole 200mg
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 16 | 16
participants
  Total number of subjects with at least 1 TEAE | 0 | 3 | 2 | 2 | 5 | 4 | 4 | 9 | 7
  Total number of subjects with at least 1 serious TEAE | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Total number of subjects with at least 1 mild TEAE | 0 | 2 | 2 | 1 | 3 | 3 | 2 | 8 | 5
  Total number of subjects with at least 1 moderate TEAE | 0 | 1 | 0 | 1 | 2 | 1 | 2 | 1 | 2
  Total number of subjects with at least 1 severe TEAE | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Total number of subjects with at least 1 treatment-related TEAE | 0 | 0 | 0 | 0 | 4 | 0 | 1 | 7 | 0
  Total number of subjects with at least 1 non treatment-related TEAE | 0 | 3 | 2 | 2 | 1 | 4 | 3 | 2 | 7

2. Secondary Outcome: AUC0-t, AUC0-inf for Voriconazole and N-oxide Voriconazole - Part 1
Description: AUC0-t = Area under the serum concentration time curve from time 0 to time t (hours) (AUC0-t) (AUC0-12 for Part 1) AUC0-inf = Area under the serum concentration time curve from time 0 to infinity
Time Frame: Part 1: at day 1 (pre-dose, at 1.5h-2h-3h-4h-12h post dose).
Population: PK Concentration Set: SAF subjects who had at least 1 quantifiable serum PK concentration recorded, analyzed according to the treatment actually taken.
Measure: Geometric Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | Part 1 - ZP-059 5mg | Part 1 - ZP-059 10mg | Part 1 - ZP-059 20mg | Part 1 - ZP-059 40mg
Number analyzed (Participants) | 6 | 6 | 6 | 6
h*ng/mL
  AUC0-t Voriconazole | 24.36 (1.45) | 73.89 (1.16) | 187.76 (1.35) | 328.37 (1.19)
  AUC0-t N-oxide Voriconazole | 298.15 (1.11) | 573.55 (1.26) | 804.24 (1.11) | 1835.81 (1.09)
  AUC0-inf Voriconazole: number analyzed (Participants) | 3 | 6 | 6 | 6
  AUC0-inf Voriconazole | 40.00 (1.00) | 78.94 (1.18) | 203.96 (1.44) | 377.19 (1.20)
  AUC0-inf N-oxide Voriconazole: number analyzed (Participants) | 6 | 5 | 4 | 3
  AUC0-inf N-oxide Voriconazole | 337.40 (1.12) | 652.99 (1.32) | 865.80 (1.07) | 1977.21 (1.11)
Statistical Analysis 1: Comparison: Part 1 - ZP-059 5mg vs Part 1 - ZP-059 10mg vs Part 1 - ZP-059 20mg vs Part 1 - ZP-059 40mg; Statistics for Voriconazole AUC0-t; Test type: Other; p < 0.0001, General power constant model; Slope = 0.62, 90% CI 2-sided [0.424 to 0.821]
Statistical Analysis 2: Comparison: Part 1 - ZP-059 5mg vs Part 1 - ZP-059 10mg vs Part 1 - ZP-059 20mg vs Part 1 - ZP-059 40mg; Statistics for Voriconazole AUC0-t; Test type: Other; p = 0.0363, General power linear model; Slope = 1.21, 90% CI 2-sided [1.050 to 1.362]
Statistical Analysis 3: Comparison: Part 1 - ZP-059 5mg vs Part 1 - ZP-059 40mg; Statistics for Voriconazole AUC0-t, 40mg vs 5mg; Test type: Other; p < 0.0001, ANOVA; Geometric mean difference = 13.48, 90% CI 2-sided [10.096 to 17.994]
Statistical Analysis 4: Comparison: Part 1 - ZP-059 5mg vs Part 1 - ZP-059 10mg vs Part 1 - ZP-059 20mg vs Part 1 - ZP-059 40mg; Statistics for N-oxide Voriconazole AUC0-t; Test type: Other; p < 0.0001, General power constant model; Slope = 1.85, 90% CI 2-sided [1.728 to 1.963]
Statistical Analysis 5: Comparison: Part 1 - ZP-059 5mg vs Part 1 - ZP-059 10mg vs Part 1 - ZP-059 20mg vs Part 1 - ZP-059 40mg; Statistics for N-oxide Voriconazole AUC0-t; Test type: Other; p = 0.0201, General power linear model; Slope = 0.87, 90% CI 2-sided [0.789 to 0.960]
Statistical Analysis 6: Comparison: Part 1 - ZP-059 5mg vs Part 1 - ZP-059 40mg; Statistics for N-oxide Voriconazole AUC0-t, 40mg vs 5mg; Test type: Other; p < 0.0001, ANOVA; Geometric mean difference = 6.16, 90% CI 2-sided [5.253 to 7.217]
Statistical Analysis 7: Comparison: Part 1 - ZP-059 5mg vs Part 1 - ZP-059 10mg vs Part 1 - ZP-059 20mg vs Part 1 - ZP-059 40mg; Statistics for Voriconazole AUC0-inf; Test type: Other; p < 0.0001, General power constant model; Slope = 0.81, 90% CI 2-sided [0.661 to 0.958]
Statistical Analysis 8: Comparison: Part 1 - ZP-059 5mg vs Part 1 - ZP-059 10mg vs Part 1 - ZP-059 20mg vs Part 1 - ZP-059 40mg; Statistics for Voriconazole AUC0-inf; Test type: Other; p = 0.1278, General power linear model; Slope = 1.12, 90% CI 2-sided [0.990 to 1.245]
Statistical Analysis 9: Comparison: Part 1 - ZP-059 5mg vs Part 1 - ZP-059 40mg; Statistics for Voriconazole AUC0-inf, 40mg vs 5mg; Test type: Other; p < 0.0001, ANOVA; Geometric mean difference = 9.43, 90% CI 2-sided [6.834 to 13.012]
Statistical Analysis 10: Comparison: Part 1 - ZP-059 5mg vs Part 1 - ZP-059 10mg vs Part 1 - ZP-059 20mg vs Part 1 - ZP-059 40mg; Statistics for N-oxide Voriconazole AUC0-inf; Test type: Other; p < 0.0001, General power constant model; Slope = 1.98, 90% CI 2-sided [1.860 to 2.106]
Statistical Analysis 11: Comparison: Part 1 - ZP-059 5mg vs Part 1 - ZP-059 10mg vs Part 1 - ZP-059 20mg vs Part 1 - ZP-059 40mg; Statistics for N-oxide Voriconazole AUC0-inf; Test type: Other; p = 0.0082, General power linear model; Slope = 0.79, 90% CI 2-sided [0.670 to 0.912]
Statistical Analysis 12: Comparison: Part 1 - ZP-059 5mg vs Part 1 - ZP-059 40mg; Statistics for N-oxide Voriconazole AUC0-inf, 40mg vs 5mg; Test type: Other; p < 0.0001, ANOVA; Geometric mean difference = 5.86, 90% CI 2-sided [4.627 to 7.421]

3. Secondary Outcome: Cmax for Voriconazole and N-oxide Voriconazole - Part 1
Description: Cmax is the highest concentration of a drug in the blood, cerebrospinal fluid, or target organ after a dose is given;
Time Frame: Part 1: at day 1 (pre-dose, at 1.5h-2h-3h-4h-12h post dose).
Population: as for outcome 2
Measure: Geometric Mean (Standard Deviation); unit: ng/mL
Arm/Group | Part 1 - ZP-059 5mg | Part 1 - ZP-059 10mg | Part 1 - ZP-059 20mg | Part 1 - ZP-059 40mg
Number analyzed (Participants) | 6 | 6 | 6 | 6
ng/mL
  Voriconazole | 8.44 (1.27) | 18.52 (1.39) | 53.37 (1.32) | 94.33 (1.18)
  N-oxide voriconazole | 57.70 (1.12) | 103.16 (1.32) | 145.79 (1.30) | 286.63 (1.15)
Statistical Analysis 1: Comparison: Part 1 - ZP-059 5mg vs Part 1 - ZP-059 10mg vs Part 1 - ZP-059 20mg vs Part 1 - ZP-059 40mg; Statistics for Voriconazole Cmax; Test type: Other; p = 0.2575, General power constant model; Slope = 0.12, 90% CI 2-sided [-0.060 to 0.308]
Statistical Analysis 2: Comparison: Part 1 - ZP-059 5mg vs Part 1 - ZP-059 10mg vs Part 1 - ZP-059 20mg vs Part 1 - ZP-059 40mg; Statistics for Voriconazole Cmax; Test type: Other; p = 0.0491, General power linear model; Slope = 1.17, 90% CI 2-sided [1.030 to 1.316]
Statistical Analysis 3: Comparison: Part 1 - ZP-059 5mg vs Part 1 - ZP-059 40mg; Statistics for Voriconazole Cmax, 40mg vs 5mg; Test type: Other; p < 0.0001, ANOVA; Geometric mean difference = 11.17, 90% CI 2-sided [8.435 to 14.803]
Statistical Analysis 4: Comparison: Part 1 - ZP-059 5mg vs Part 1 - ZP-059 10mg vs Part 1 - ZP-059 20mg vs Part 1 - ZP-059 40mg; Statistics for N-oxide Voriconazole Cmax; Test type: Other; p < 0.0001, General power constant model; Slope = 1.25, 90% CI 2-sided [1.135 to 1.363]
Statistical Analysis 5: Comparison: Part 1 - ZP-059 5mg vs Part 1 - ZP-059 10mg vs Part 1 - ZP-059 20mg vs Part 1 - ZP-059 40mg; Statistics for N-oxide Voriconazole Cmax; Test type: Other; p = 0.0003, General power linear model; Slope = 0.74, 90% CI 2-sided [0.634 to 0.843]
Statistical Analysis 6: Comparison: Part 1 - ZP-059 5mg vs Part 1 - ZP-059 40mg; Statistics for N-oxide Voriconazole Cmax, 40mg vs 5mg; Test type: Other; p < 0.0001, ANOVA; Geometric mean difference = 4.97, 90% CI 2-sided [3.946 to 6.254]

4. Secondary Outcome: Tmax and T1/2 for Voriconazole and N-oxide Voriconazole - Part 1
Description: Tmax= Time to maximum concentration (Cmax). T 1/2 = Elimination half-life: the time taken for the plasma concentration to fall by half its original value.
Time Frame: Part 1: at day 1 (pre-dose, at 1.5h-2h-3h-4h-12h post dose).
Population: as for outcome 2
Measure: Geometric Mean (Standard Deviation); unit: hours
Arm/Group | Part 1 - ZP-059 5mg | Part 1 - ZP-059 10mg | Part 1 - ZP-059 20mg | Part 1 - ZP-059 40mg
Number analyzed (Participants) | 6 | 6 | 6 | 6
hours
  Tmax Voriconazole | 1.57 (1.11) | 1.50 (1.00) | 1.50 (1.00) | 1.50 (1.00)
  Tmax N-oxide voriconazole | 1.57 (1.11) | 1.50 (1.00) | 1.85 (1.29) | 1.65 (1.15)
  T1/2 Voriconazole: number analyzed (Participants) | 4 | 6 | 6 | 6
  T1/2 Voriconazole | 2.67 (1.42) | 3.07 (1.09) | 3.20 (1.17) | 3.63 (1.22)
  T1/2 N-oxide voriconazole: number analyzed (Participants) | 6 | 6 | 5 | 6
  T1/2 N-oxide voriconazole | 3.60 (1.08) | 3.59 (1.21) | 3.38 (1.27) | 4.43 (1.26)

5. Secondary Outcome: Kel for Voriconazole and N-oxide Voriconazole - Part 1
Description: Kel (Elimination rate constant): is a value used to describe the rate at which a drug is removed from the human system.
  It is equivalent to the fraction of a substance that is removed per unit time measured at any particular instant and has units of 1/h.
Time Frame: Part 1: at day 1 (pre-dose, at 1.5h-2h-3h-4h-12h post dose).
Population: as for outcome 2
Measure: Geometric Mean (Standard Deviation); unit: 1/h
Arm/Group | Part 1 - ZP-059 5mg | Part 1 - ZP-059 10mg | Part 1 - ZP-059 20mg | Part 1 - ZP-059 40mg
Number analyzed (Participants) | 6 | 6 | 6 | 6
1/h
  Voriconazole: number analyzed (Participants) | 5 | 6 | 6 | 6
  Voriconazole | 0.30 (1.52) | 0.23 (1.09) | 0.22 (1.17) | 0.19 (1.22)
  N-oxide voriconazole: number analyzed (Participants) | 6 | 6 | 5 | 6
  N-oxide voriconazole | 0.19 (1.08) | 0.19 (1.21) | 0.20 (1.27) | 0.16 (1.26)

6. Secondary Outcome: CL/F for Voriconazole - Part 1
Description: Apparent clearance: Equal to the drug dose divided by the area-under-the-curve; is an important pharmacokinetic parameter and plays an important role in the selection of a safe and tolerable dose for first-in-human studies.
Time Frame: Part 1: at day 1 (pre-dose, at 1.5h-2h-3h-4h-12h post dose).
Population: as for outcome 2
Measure: Geometric Mean (Standard Deviation); unit: L/h
Arm/Group | Part 1 - ZP-059 5mg | Part 1 - ZP-059 10mg | Part 1 - ZP-059 20mg | Part 1 - ZP-059 40mg
Number analyzed (Participants) | 6 | 6 | 6 | 6
L/h | 131.2 (1.04) | 124.6 (1.17) | 97.7 (1.39) | 108.7 (1.22)

7. Secondary Outcome: Vz/F for Voriconazole - Part 1
Description: Vz/F=Apparent volume of distribution during terminal phase.
Time Frame: Part 1: at day 1 (pre-dose, at 1.5h-2h-3h-4h-12h post dose).
Population: as for outcome 2
Measure: Geometric Mean (Standard Deviation); unit: liters
Arm/Group | Part 1 - ZP-059 5mg | Part 1 - ZP-059 10mg | Part 1 - ZP-059 20mg | Part 1 - ZP-059 40mg
Number analyzed (Participants) | 3 | 6 | 6 | 6
liters | 614.3 (1.09) | 553.1 (1.14) | 450.9 (1.25) | 569.6 (1.20)

8. Secondary Outcome: MR AUC0-t, MR AUC0-inf for N-oxide Voriconazole - Part 1
Description: MR = metabolite ratio. Metabolite ratios (as appropriate) will be calculated for AUC and Cmax parameters.
  Area under the serum concentration time curve from time 0 to time t (hours) (AUC0-t)
Time Frame: Part 1: at day 1 (pre-dose, at 1.5h-2h-3h-4h-12h post dose).
Population: as for outcome 2
Measure: Geometric Mean (Standard Deviation); unit: ratio
Arm/Group | Part 1 - ZP-059 5mg | Part 1 - ZP-059 10mg | Part 1 - ZP-059 20mg | Part 1 - ZP-059 40mg
Number analyzed (Participants) | 6 | 6 | 6 | 6
ratio
  MR AUC0-t | 12.25 (1.36) | 7.76 (1.40) | 4.28 (1.43) | 5.59 (1.14)
  MR AUC0-inf: number analyzed (Participants) | 5 | 6 | 5 | 6
  MR AUC0-inf | 10.92 (1.20) | 8.18 (1.39) | 4.92 (1.42) | 6.12 (1.08)

9. Secondary Outcome: MR Cmax for N-oxide Voriconazole - Part 1
Description: MR = metabolite ratio. Metabolite ratios (as appropriate) will be calculated for AUC and Cmax parameters.
  Cmax is the highest concentration of a drug in the blood, cerebrospinal fluid, or target organ after a dose is given.
Time Frame: Part 1: at day 1 (pre-dose, at 1.5h-2h-3h-4h-12h post dose).
Population: as for outcome 2
Measure: Geometric Mean (Standard Deviation); unit: ratio
Arm/Group | Part 1 - ZP-059 5mg | Part 1 - ZP-059 10mg | Part 1 - ZP-059 20mg | Part 1 - ZP-059 40mg
Number analyzed (Participants) | 6 | 6 | 6 | 6
ratio | 6.84 (1.27) | 5.57 (1.73) | 2.73 (1.51) | 3.04 (1.31)

10. Secondary Outcome: AUC0-t, AUC0-inf for Voriconazole and N-oxide Voriconazole - Part 2
Description: AUC0-t = Area under the serum concentration time curve from time 0 to time t (hours) (AUC0-t) (AUC0-24 for Part 2) AUC0-inf = Area under the serum concentration time curve from time 0 to infinity
Time Frame: Part 2: Day 1 (1.5, 2, 3, 4, and 12 hours post-0-hour dose) and Day 10 (post-0-hour dose at 1.5, 2, 3, 4, and 12 hours)
Population: as for outcome 2
Measure: Geometric Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | Part 2 - ZP-059 10mg Bid | Part 2 - ZP-059 20mg Bid | Part 2 - ZP-059 40mg qd
Number analyzed (Participants) | 6 | 6 | 6
h*ng/mL
  AUC0-t Voriconazole - Day 1 | 69.65 (1.39) | 139.29 (1.21) | 329.28 (1.19)
  AUC0-inf Voriconazole - Day 1: number analyzed (Participants) | 5 | 6 | 6
  AUC0-inf Voriconazole - Day 1 | 78.20 (1.40) | 155.72 (1.16) | 358.13 (1.20)
  AUC0-t Voriconazole - Day 10 | 91.00 (1.36) | 256.04 (1.41) | 480.22 (1.27)
  AUC0-inf Voriconazole - Day 10: number analyzed (Participants) | 6 | 5 | 6
  AUC0-inf Voriconazole - Day 10 | 97.78 (1.35) | 258.66 (1.44) | 493.04 (1.29)
  AUC0-t N-oxide Voriconazole - Day 1 | 391.28 (1.19) | 769.65 (1.15) | 1990.76 (1.23)
  AUC0-inf N-oxide Voriconazole - Day 1: number analyzed (Participants) | 6 | 6 | 4
  AUC0-inf N-oxide Voriconazole - Day 1 | 439.14 (1.20) | 849.27 (1.17) | 2001.85 (1.24)
  AUC0-t N-oxide Voriconazole - Day 10 | 728.68 (1.31) | 1784.63 (1.40) | 3353.43 (1.27)
  AUC0-inf N-oxide Voriconazole - Day 10: number analyzed (Participants) | 6 | 5 | 5
  AUC0-inf N-oxide Voriconazole - Day 10 | 752.99 (1.32) | 1807.93 (1.47) | 3174.66 (1.19)
Statistical Analysis 1: Comparison: Part 2 - ZP-059 10mg Bid vs Part 2 - ZP-059 20mg Bid; Statistics for Voriconazole AUC0-t Day 1; Test type: Other; p = 0.0004, ANOVA; Slope = 2.00, 90% CI 2-sided [1.528 to 2.617]
Statistical Analysis 2: Comparison: Part 2 - ZP-059 10mg Bid vs Part 2 - ZP-059 40mg qd; Statistics for Voriconazole AUC0-t Day 1; Test type: Other; p < 0.0001, ANOVA; Slope = 4.73, 90% CI 2-sided [3.612 to 6.187]
Statistical Analysis 3: Comparison: Part 2 - ZP-059 10mg Bid vs Part 2 - ZP-059 20mg Bid; Statistics for Voriconazole AUC0-t day 10; Test type: Other; p < 0.0001, ANOVA; Slope = 2.81, 90% CI 2-sided [2.017 to 3.925]
Statistical Analysis 4: Comparison: Part 2 - ZP-059 10mg Bid vs Part 2 - ZP-059 40mg qd; Statistics for Voriconazole AUC0-t Day 10; Test type: Other; p < 0.0001, ANOVA; Slope = 5.28, 90% CI 2-sided [3.783 to 7.361]
Statistical Analysis 5: Comparison: Part 2 - ZP-059 10mg Bid vs Part 2 - ZP-059 20mg Bid; Statistics for N-oxide Voriconazole AUC0-t Day 1; Test type: Other; p < 0.0001, ANOVA; Slope = 1.97, 90% CI 2-sided [1.615 to 2.396]
Statistical Analysis 6: Comparison: Part 2 - ZP-059 10mg Bid vs Part 2 - ZP-059 40mg qd; Statistics for N-oxide Voriconazole AUC0-t Day 1; Test type: Other; p < 0.0001, ANOVA; Slope = 5.09, 90% CI 2-sided [4.178 to 6.196]
Statistical Analysis 7: Comparison: Part 2 - ZP-059 10mg Bid vs Part 2 - ZP-059 20mg Bid; Statistics for N-oxide Voriconazole AUC0-t Day 10; Test type: Other; p = 0.0002, ANOVA; Slope = 2.45, 90% CI 2-sided [1.791 to 3.349]
Statistical Analysis 8: Comparison: Part 2 - ZP-059 10mg Bid vs Part 2 - ZP-059 40mg qd; Statistics for N-oxide Voriconazole AUC0-t Day 10; Test type: Other; p < 0.0001, ANOVA; Slope = 4.60, 90% CI 2-sided [3.365 to 6.294]
Statistical Analysis 9: Comparison: Part 2 - ZP-059 10mg Bid vs Part 2 - ZP-059 20mg Bid; Statistics for Voriconazole AUC0-inf Day 1; Test type: Other; p = 0.0005, ANOVA; Slope = 1.99, 90% CI 2-sided [1.524 to 2.602]
Statistical Analysis 10: Comparison: Part 2 - ZP-059 10mg Bid vs Part 2 - ZP-059 40mg qd; Statistics for Voriconazole AUC0-inf Day 1; Test type: Other; p < 0.0001, ANOVA; Slope = 4.58, 90% CI 2-sided [3.505 to 5.984]
Statistical Analysis 11: Comparison: Part 2 - ZP-059 10mg Bid vs Part 2 - ZP-059 20mg Bid; Statistics for Voriconazole AUC0-inf Day 10; Test type: Other; p = 0.0003, ANOVA; Slope = 2.65, 90% CI 2-sided [1.851 to 3.781]
Statistical Analysis 12: Comparison: Part 2 - ZP-059 10mg Bid vs Part 2 - ZP-059 40mg qd; Statistics for Voriconazole AUC0-inf Day 10; Test type: Other; p < 0.0001, ANOVA; Slope = 5.04, 90% CI 2-sided [3.587 to 7.088]
Statistical Analysis 13: Comparison: Part 2 - ZP-059 10mg Bid vs Part 2 - ZP-059 20mg Bid; Statistics for N-oxide Voriconazole AUC0-inf Day 1; Test type: Other; p < 0.0001, ANOVA; Slope = 1.93, 90% CI 2-sided [1.569 to 2.384]
Statistical Analysis 14: Comparison: Part 2 - ZP-059 10mg Bid vs Part 2 - ZP-059 40mg qd; Statistics for N-oxide Voriconazole AUC0-inf Day 1; Test type: Other; p < 0.0001, ANOVA; Slope = 4.56, 90% CI 2-sided [3.608 to 5.759]
Statistical Analysis 15: Comparison: Part 2 - ZP-059 10mg Bid vs Part 2 - ZP-059 20mg Bid; Statistics for N-oxide Voriconazole AUC0-inf Day 10; Test type: Other; p = 0.0007, ANOVA; Slope = 2.40, 90% CI 2-sided [1.694 to 3.402]
Statistical Analysis 16: Comparison: Part 2 - ZP-059 10mg Bid vs Part 2 - ZP-059 40mg qd; Statistics for N-oxide Voriconazole AUC0-inf Day 10; Test type: Other; p < 0.0001, ANOVA; Slope = 4.22, 90% CI 2-sided [2.975 to 5.974]

11. Secondary Outcome: Cmax for Voriconazole and N-oxide Voriconazole - Part 2
Description: Cmax is the highest concentration of a drug in the blood, cerebrospinal fluid, or target organ after a dose is given;
Time Frame: Part 2: Day 1 (1.5, 2, 3, 4, and 12 hours post-0-hour dose) and Day 10 (post-0-hour dose at 1.5, 2, 3, 4, and 12 hours)
Population: as for outcome 2
Measure: Geometric Mean (Standard Deviation); unit: ng/mL
Arm/Group | Part 2 - ZP-059 10mg Bid | Part 2 - ZP-059 20mg Bid | Part 2 - ZP-059 40mg qd
Number analyzed (Participants) | 6 | 6 | 6
ng/mL
  Voriconazole - Day 1 | 19.87 (1.29) | 40.42 (1.33) | 96.77 (1.16)
  Voriconazole - Day 10 | 21.38 (1.21) | 57.11 (1.33) | 127.54 (1.20)
  N-oxide Voriconazole - Day 1 | 71.66 (1.24) | 144.43 (1.11) | 339.11 (1.15)
  N-oxide Voriconazole - Day 10 | 102.78 (1.30) | 217.76 (1.23) | 412.40 (1.21)
Statistical Analysis 1: Comparison: Part 2 - ZP-059 10mg Bid vs Part 2 - ZP-059 20mg Bid; Statistics for Voriconazole Cmax Day 1; Test type: Other; p = 0.0003, ANOVA; Slope = 2.03, 90% CI 2-sided [1.562 to 2.650]
Statistical Analysis 2: Comparison: Part 2 - ZP-059 10mg Bid vs Part 2 - ZP-059 40mg qd; Statistics for Voriconazole Cmax Day 1; Test type: Other; p < 0.0001, ANOVA; Slope = 4.87, 90% CI 2-sided [3.740 to 6.345]
Statistical Analysis 3: Comparison: Part 2 - ZP-059 10mg Bid vs Part 2 - ZP-059 20mg Bid; Statistics for Voriconazole Cmax Day 10; Test type: Other; p < 0.0001, ANOVA; Slope = 2.67, 90% CI 2-sided [2.081 to 3.429]
Statistical Analysis 4: Comparison: Part 2 - ZP-059 10mg Bid vs Part 2 - ZP-059 40mg qd; Statistics for Voriconazole Cmax Day 10; Test type: Other; p < 0.0001, ANOVA; Slope = 5.97, 90% CI 2-sided [4.647 to 7.658]
Statistical Analysis 5: Comparison: Part 2 - ZP-059 10mg Bid vs Part 2 - ZP-059 20mg Bid; Statistics for N-oxide Voriconazole Cmax Day 1; Test type: Other; p < 0.0001, ANOVA; Slope = 2.02, 90% CI 2-sided [1.688 to 2.406]
Statistical Analysis 6: Comparison: Part 2 - ZP-059 10mg Bid vs Part 2 - ZP-059 40mg qd; Statistics for N-oxide Voriconazole Cmax Day 1; Test type: Other; p < 0.0001, ANOVA; Slope = 4.73, 90% CI 2-sided [3.964 to 5.650]
Statistical Analysis 7: Comparison: Part 2 - ZP-059 10mg Bid vs Part 2 - ZP-059 20mg Bid; Statistics for N-oxide Voriconazole Cmax Day 10; Test type: Other; p < 0.0001, ANOVA; Slope = 2.12, 90% CI 2-sided [1.655 to 2.711]
Statistical Analysis 8: Comparison: Part 2 - ZP-059 10mg Bid vs Part 2 - ZP-059 40mg qd; Statistics for N-oxide Voriconazole Cmax day 10; Test type: Other; p < 0.0001, ANOVA; Slope = 4.01, 90% CI 2-sided [3.135 to 5.135]

12. Secondary Outcome: Tmax and T1/2 for Voriconazole and N-oxide Voriconazole - Part 2
Description: as for outcome 4
Time Frame: Part 2: Day 1 (1.5, 2, 3, 4, and 12 hours post-0-hour dose) and Day 10 (post-0-hour dose at 1.5, 2, 3, 4, and 12 hours)
Population: as for outcome 2
Measure: Geometric Mean (Standard Deviation); unit: hours
Arm/Group | Part 2 - ZP-059 10mg Bid | Part 2 - ZP-059 20mg Bid | Part 2 - ZP-059 40mg qd
Number analyzed (Participants) | 6 | 6 | 6
hours
  Tmax Voriconazole - Day 1 | 1.50 (1.00) | 1.50 (1.00) | 1.57 (1.11)
  Tmax Voriconazole - Day 10 | 1.50 (1.00) | 1.50 (1.00) | 1.50 (1.00)
  Tmax N-oxide Voriconazole - Day 1 | 1.65 (1.15) | 1.50 (1.00) | 1.65 (1.15)
  Tmax N-oxide Voriconazole - Day 10 | 1.57 (1.11) | 1.57 (1.11) | 2.33 (1.45)
  T1/2 Voriconazole - Day 1 | 3.60 (1.36) | 3.53 (1.25) | 3.24 (1.08)
  T1/2 Voriconazole - Day 10: number analyzed (Participants) | 6 | 5 | 6
  T1/2 Voriconazole - Day 10 | 4.40 (1.41) | 5.15 (1.29) | 4.48 (1.15)
  T1/2 N-oxide Voriconazole - Day 1 | 3.45 (1.08) | 3.20 (1.11) | 3.82 (1.44)
  T1/2 N-oxide Voriconazole - Day 10: number analyzed (Participants) | 6 | 5 | 5
  T1/2 N-oxide Voriconazole - Day 10 | 4.52 (1.16) | 5.04 (1.24) | 4.14 (1.21)

13. Secondary Outcome: Kel for Voriconazole and N-oxide Voriconazole - Part 2
Description: as for outcome 5
Time Frame: Part 2: Day 1 (1.5, 2, 3, 4, and 12 hours post-0-hour dose) and Day 10 (post-0-hour dose at 1.5, 2, 3, 4, and 12 hours)
Population: as for outcome 2
Measure: Geometric Mean (Standard Deviation); unit: 1/h
Arm/Group | Part 2 - ZP-059 10mg Bid | Part 2 - ZP-059 20mg Bid | Part 2 - ZP-059 40mg qd
Number analyzed (Participants) | 6 | 6 | 6
1/h
  Voriconazole - Day 1 | 0.19 (1.35) | 0.20 (1.25) | 0.21 (1.08)
  Voriconazole - Day 10: number analyzed (Participants) | 6 | 5 | 6
  Voriconazole - Day 10 | 0.16 (1.41) | 0.13 (1.29) | 0.15 (1.15)
  N-oxide Voriconazole - Day 1 | 0.20 (1.08) | 0.22 (1.11) | 0.18 (1.44)
  N-oxide Voriconazole - Day 10: number analyzed (Participants) | 6 | 5 | 5
  N-oxide Voriconazole - Day 10 | 0.15 (1.16) | 0.14 (1.24) | 0.17 (1.21)

14. Secondary Outcome: CL/F for Voriconazole - Part 2
Description: as for outcome 6
Time Frame: Part 2: Only at Day 10 (post-0-hour dose at 1.5, 2, 3, 4, and 12 hours)
Population: as for outcome 2
Measure: Geometric Mean (Standard Deviation); unit: L/h
Arm/Group | Part 2 - ZP-059 10mg Bid | Part 2 - ZP-059 20mg Bid | Part 2 - ZP-059 40mg qd
Number analyzed (Participants) | 6 | 6 | 6
L/h | 120.9 (1.29) | 93.1 (1.32) | 93.5 (1.25)

15. Secondary Outcome: Swing for Voriconazole and N-oxide Voriconazole - Part 2
Description: Swing for voriconazole and N-oxide voriconazole = [(Cmax - Cmin) / Cmin]*100%
Time Frame: Part 2: Only at Day 10 (post-0-hour dose at 1.5, 2, 3, 4, and 12 hours)
Population: as for outcome 2
Measure: Geometric Mean (Standard Deviation); unit: percentage concentration
Arm/Group | Part 2 - ZP-059 10mg Bid | Part 2 - ZP-059 20mg Bid | Part 2 - ZP-059 40mg qd
Number analyzed (Participants) | 6 | 6 | 6
percentage concentration
  Voriconazole | 10.50 (1.48) | 9.62 (1.68) | 55.16 (1.63)
  N-oxide Voriconazole | 4.60 (1.16) | 3.81 (1.48) | 20.65 (2.70)

16. Secondary Outcome: AUCtau for Voriconazole and N-oxide Voriconazole - Part 2
Description: Area under the serum concentration time curve for the dosing interval
Time Frame: Part 2: Only at Day 10 (post-0-hour dose at 1.5, 2, 3, 4, and 12 hours)
Population: as for outcome 2
Measure: Geometric Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | Part 2 - ZP-059 10mg Bid | Part 2 - ZP-059 20mg Bid | Part 2 - ZP-059 40mg qd
Number analyzed (Participants) | 6 | 6 | 6
h*ng/mL
  Voriconazole | 82.82 (1.30) | 215.56 (1.32) | 427.57 (1.25)
  N-oxide Voriconazole | 620.89 (1.28) | 1438.74 (1.31) | 2803.51 (1.20)

17. Secondary Outcome: Css,av for Voriconazole and N-oxide Voriconazole - Part 2
Description: Css,av or Css(ave): Average drug concentration at steady state; Steady-state concentration (Css) occurs when the amount of a drug being absorbed is the same amount that's being cleared from the body when the drug is given continuously or repeatedly
Time Frame: Part 2: Only at Day 10 (post-0-hour dose at 1.5, 2, 3, 4, and 12 hours)
Population: as for outcome 2
Measure: Geometric Mean (Standard Deviation); unit: ng/mL
Arm/Group | Part 2 - ZP-059 10mg Bid | Part 2 - ZP-059 20mg Bid | Part 2 - ZP-059 40mg qd
Number analyzed (Participants) | 6 | 6 | 6
ng/mL
  Voriconazole | 6.91 (1.30) | 17.95 (1.32) | 35.64 (1.25)
  N-oxide Voriconazole | 51.75 (1.28) | 119.88 (1.31) | 233.63 (1.20)

18. Secondary Outcome: Fluctuation for Voriconazole and N-oxide Voriconazole - Part 2
Description: Peak trough fluctuation in serum concentrations within one dosing interval at steady state. Fluctuation - Over the Dosing Interval - is expressed as percentage concentration.
Time Frame: Part 2: Only at Day 10 (post-0-hour dose at 1.5, 2, 3, 4, and 12 hours)
Population: as for outcome 2
Measure: Geometric Mean (Standard Deviation); unit: percentage concentration
Arm/Group | Part 2 - ZP-059 10mg Bid | Part 2 - ZP-059 20mg Bid | Part 2 - ZP-059 40mg qd
Number analyzed (Participants) | 6 | 6 | 6
percentage concentration
  Voriconazole | 281.0 (1.15) | 284.9 (1.24) | 350.8 (1.10)
  N-oxide Voriconazole | 162.8 (1.08) | 141.8 (1.21) | 163.8 (1.30)

19. Secondary Outcome: Rac for Voriconazole and N-oxide Voriconazole - Part 2
Description: Accumulation ratio. The drug accumulation ratio (Rac) is the ratio of accumulation of a drug under steady state conditions as compared to a single dose. The higher the value, the more the drug accumulates in the body. An Rac of 1 means no accumulation.
Time Frame: Part 2: Only at Day 10 (post-0-hour dose at 1.5, 2, 3, 4, and 12 hours)
Population: as for outcome 2
Measure: Geometric Mean (Standard Deviation); unit: ratio
Arm/Group | Part 2 - ZP-059 10mg Bid | Part 2 - ZP-059 20mg Bid | Part 2 - ZP-059 40mg qd
Number analyzed (Participants) | 6 | 6 | 6
ratio
  Voriconazole | 1.19 (1.17) | 1.55 (1.29) | 1.30 (1.27)
  N-oxide Voriconazole | 1.59 (1.11) | 1.87 (1.20) | 1.41 (1.10)

20. Secondary Outcome: Rlinear for Voriconazole and N-oxide Voriconazole - Part 2
Description: Rlinear means linearity ratio for Area Under the Serum Concentration-Time Curve from time zero to infinity.
Time Frame: Part 2: Only at Day 10 (post-0-hour dose at 1.5, 2, 3, 4, and 12 hours)
Population: as for outcome 2
Measure: Geometric Mean (Standard Deviation); unit: ratio
Arm/Group | Part 2 - ZP-059 10mg Bid | Part 2 - ZP-059 20mg Bid | Part 2 - ZP-059 40mg qd
Number analyzed (Participants) | 6 | 6 | 6
ratio
  Voriconazole: number analyzed (Participants) | 5 | 6 | 6
  Voriconazole | 1.06 (1.14) | 1.38 (1.25) | 1.19 (1.26)
  N-oxide Voriconazole: number analyzed (Participants) | 6 | 5 | 4
  N-oxide Voriconazole | 1.42 (1.12) | 1.70 (1.21) | 1.30 (1.17)

21. Secondary Outcome: MR AUC0-t, MR AUC0-inf and MR AUCtau for N-oxide Voriconazole - Part 2
Description: as for outcome 8
Time Frame: Part 2: Day 1 (1.5, 2, 3, 4, and 12 hours post-0-hour dose) and Day 10 (post-0-hour dose at 1.5, 2, 3, 4, and 12 hours)
Population: as for outcome 2
Measure: Geometric Mean (Standard Deviation); unit: ratio
Arm/Group | Part 2 - ZP-059 10mg Bid | Part 2 - ZP-059 20mg Bid | Part 2 - ZP-059 40mg qd
Number analyzed (Participants) | 6 | 6 | 6
ratio
  MR AUC0-t N-oxide Voriconazole - Day 1 | 5.62 (1.50) | 5.53 (1.32) | 6.04 (1.27)
  MR AUC0-inf N-oxide Voriconazole - Day 1: number analyzed (Participants) | 5 | 6 | 4
  MR AUC0-inf N-oxide Voriconazole - Day 1 | 5.68 (1.52) | 5.45 (1.29) | 5.55 (1.20)
  MR AUC0-t N-oxide Voriconazole - Day 10 | 8.01 (1.40) | 6.97 (1.32) | 6.98 (1.16)
  MR AUC0-inf N-oxide Voriconazole - Day 10: number analyzed (Participants) | 6 | 5 | 5
  MR AUC0-inf N-oxide Voriconazole - Day 10 | 7.70 (1.40) | 6.99 (1.34) | 7.11 (1.18)
  MR AUCtau N-oxide Voriconazole - Day 10 | 7.50 (1.39) | 6.68 (1.30) | 6.56 (1.20)

22. Secondary Outcome: MR Cmax N-oxide Voriconazole - Part 2
Description: as for outcome 9
Time Frame: Part 2: Day 1 (1.5, 2, 3, 4, and 12 hours post-0-hour dose) and Day 10 (post-0-hour dose at 1.5, 2, 3, 4, and 12 hours)
Population: as for outcome 2
Measure: Geometric Mean (Standard Deviation); unit: ratio
Arm/Group | Part 2 - ZP-059 10mg Bid | Part 2 - ZP-059 20mg Bid | Part 2 - ZP-059 40mg qd
Number analyzed (Participants) | 6 | 6 | 6
ratio
  N-oxide Voriconazole - Day 1 | 3.61 (1.50) | 3.57 (1.40) | 3.50 (1.22)
  N-oxide Voriconazole - Day 10 | 4.81 (1.38) | 3.81 (1.34) | 3.23 (1.37)

23. Secondary Outcome: Cmax for Voriconazole and N-oxide Voriconazole - Part 3
Description: Cmax is the highest concentration of a drug in the blood, cerebrospinal fluid, or target organ after a dose is given;
Time Frame: Day 1 of the respective treatment period 1 or 2
Population: as for outcome 2
Measure: Geometric Mean (Standard Deviation); unit: ng/mL
Groups:
- Part 3 - ZP-059: Crossover treatment period: Single inhaled dose (20 mg) of ZP-059 5mg capsules administered via DPI, and a single dose of oral voriconazole (200 mg Vfend® tablet) on the morning of Day 1 of the respective treatment period with a washout period of at least 96 hours.
  Voriconazole inhaled: Part 1 (SAD): eligible subjects received a single ascending inhaled dose (5 mg, 10 mg, 20 mg, and 40 mg) of ZP-059 5mg capsules administered via dry powder inhaler (DPI) on the morning of Day 1.
  Part 2 (MAD): eligible subjects received 2 (10mg twice daily [BID]) or 4 [20mg BID]) inhaled doses of ZP-059 5mg capsules administered via DPI BID for 9 days and once in the morning of Day 10, or 8 inhaled doses of ZP-059 5 mg capsules (40mg once daily [QD]) for 10 days. For QD dosing, subjects received QD doses of ZP-059 (at hour 0) on Days 1 to 10.
  Part 3 (2-period crossover): eligible subjects received a single inhaled dose (20mg) of ZP-059 5mg capsules administered via DPI on the morning of Day 1 according to the crossover scheme of the study.
  ZP-059 (inhaled voriconazole) was provided in clear, colorless size 3 hydroxypropylmethylcellulose hard capsules, which were individually and manually triggered by a breath actuated inhalation device (RS01 monodose inhaler).
  oral voriconazole: Part 3 (2-period crossover): eligible subjects received a single dose of oral voriconazole (200mg oral film-coated tablet, Vfend) on the morning of Day 1 according to the crossover scheme of the study.
- Part 3 - Oral Voriconazole: Crossover treatment period: Single dose of oral voriconazole (200 mg Vfend® tablet), and a single inhaled dose (20 mg) of ZP-059 5mg capsules administered via DPI on the morning of Day 1 of the respective treatment period with a washout period of at least 96 hours.
  Voriconazole inhaled: Part 1 (SAD): eligible subjects received a single ascending inhaled dose (5 mg, 10 mg, 20 mg, and 40 mg) of ZP-059 5mg capsules administered via dry powder inhaler (DPI) on the morning of Day 1.
  Part 2 (MAD): eligible subjects received 2 (10mg twice daily [BID]) or 4 [20mg BID]) inhaled doses of ZP-059 5mg capsules administered via DPI BID for 9 days and once in the morning of Day 10, or 8 inhaled doses of ZP-059 5 mg capsules (40mg once daily [QD]) for 10 days. For QD dosing, subjects received QD doses of ZP-059 (at hour 0) on Days 1 to 10.
  Part 3 (2-period crossover): eligible subjects received a single inhaled dose (20mg) of ZP-059 5mg capsules administered via DPI on the morning of Day 1 according to the crossover scheme of the study.
  ZP-059 (inhaled voriconazole) was provided in clear, colorless size 3 hydroxypropylmethylcellulose hard capsules, which were individually and manually triggered by a breath actuated inhalation device (RS01 monodose inhaler).
  oral voriconazole: Part 3 (2-period crossover): eligible subjects received a single dose of oral voriconazole (200mg oral film-coated tablet, Vfend) on the morning of Day 1 according to the crossover scheme of the study.
Arm/Group | Part 3 - ZP-059 | Part 3 - Oral Voriconazole
Number analyzed (Participants) | 16 | 16
ng/mL
  Voriconazole | 108.08 (1.42) | 863.22 (1.44)
  N-oxide Voriconazole | 151.43 (1.25) | 1589.05 (1.25)

24. Secondary Outcome: Vz/F for Voriconazole - Part 3
Description: Vz/F=Apparent volume of distribution during terminal phase.
Time Frame: Only at Day 10
Population: as for outcome 2
Measure: Geometric Mean (Standard Deviation); unit: Liters
Arm/Group | Part 2 - ZP-059 10mg Bid | Part 2 - ZP-059 20mg Bid | Part 2 - ZP-059 40mg qd
Number analyzed (Participants) | 6 | 5 | 6
Liters | 767.1 (1.47) | 714.3 (1.25) | 604.9 (1.13)

25. Secondary Outcome: AUC0-t, AUC0-inf for Voriconazole and N-oxide Voriconazole - Part 3
Description: AUC0-t = Area under the serum concentration time curve from time 0 to time t (hours) (AUC0-t) (AUC0-96 for Part 3) AUC0-inf = Area under the serum concentration time curve from time 0 to infinity
Time Frame: Day 1 of the respective treatment period 1 or 2
Population: as for outcome 2
Measure: Geometric Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | Part 3 - ZP-059 | Part 3 - Oral Voriconazole
Number analyzed (Participants) | 16 | 16
h*ng/mL
  AUC0-t Voriconazole | 290.02 (1.87) | 3726.68 (1.91)
  AUC0-inf Voriconazole: number analyzed (Participants) | 15 | 16
  AUC0-inf Voriconazole | 269.61 (1.56) | 3800.41 (1.92)
  AUC0-t N-oxide Voriconazole | 1128.69 (1.27) | 21504.52 (1.20)
  AUC0-inf N-oxide Voriconazole | 1154.35 (1.26) | 21788.46 (1.20)

26. Secondary Outcome: Tmax and T1/2 for Voriconazole and N-oxide Voriconazole - Part 3
Description: as for outcome 4
Time Frame: Day 1 of the respective treatment period 1 or 2 (Pre-dose, 0.25h, 0.75h 1.5h, 2h ,3h ,4h ,6h ,8h ,12h ,16h , 24h ,48h after dosing)
Population: as for outcome 2
Measure: Geometric Mean (Standard Deviation); unit: hours
Arm/Group | Part 3 - ZP-059 | Part 3 - Oral Voriconazole
Number analyzed (Participants) | 16 | 16
hours
  Tmax Voriconazole | 0.43 (3.64) | 1.16 (1.40)
  Tmax N-oxide Voriconazole | 1.74 (1.31) | 2.76 (1.52)
  T1/2 Voriconazole: number analyzed (Participants) | 15 | 16
  T1/2 Voriconazole | 5.13 (1.27) | 6.93 (1.32)
  T1/2 N-oxide Voriconazole | 4.68 (1.19) | 6.42 (1.35)

27. Secondary Outcome: CL/F for Voriconazole - Part 3
Description: as for outcome 6
Time Frame: Day 1 of the respective treatment period 1 or 2
Population: as for outcome 2
Measure: Geometric Mean (Standard Deviation); unit: L/h
Arm/Group | Part 3 - ZP-059 | Part 3 - Oral Voriconazole
Number analyzed (Participants) | 15 | 16
L/h | 74.2 (1.57) | 52.4 (1.93)

28. Secondary Outcome: Kel for Voriconazole and N-oxide Voriconazole - Part 3
Description: as for outcome 5
Time Frame: Day 1 of the respective treatment period 1 or 2
Population: as for outcome 2
Measure: Geometric Mean (Standard Deviation); unit: 1/h
Arm/Group | Part 3 - ZP-059 | Part 3 - Oral Voriconazole
Number analyzed (Participants) | 16 | 16
1/h
  Voriconazole: number analyzed (Participants) | 15 | 16
  Voriconazole | 0.14 (1.26) | 0.10 (1.31)
  N-oxide Voriconazole | 0.15 (1.19) | 0.11 (1.34)

29. Secondary Outcome: Vz/F for Voriconazole - Part 3
Description: Vz/F=Apparent volume of distribution during terminal phase.
Time Frame: Day 1 of the respective treatment period 1 or 2
Population: as for outcome 2
Measure: Geometric Mean (Standard Deviation); unit: Liters
Arm/Group | Part 3 - ZP-059 | Part 3 - Oral Voriconazole
Number analyzed (Participants) | 15 | 16
Liters | 549.0 (1.46) | 526.0 (1.69)

30. Secondary Outcome: MR AUC0-t and MR AUC0-inf for N-oxide Voriconazole - Part 3
Description: as for outcome 8
Time Frame: Day 1 of the respective treatment period 1 or 2
Population: as for outcome 2
Measure: Geometric Mean (Standard Deviation); unit: ratio
Arm/Group | Part 3 - ZP-059 | Part 3 - Oral Voriconazole
Number analyzed (Participants) | 16 | 16
ratio
  MR AUC0-t | 3.89 (1.92) | 5.77 (1.81)
  MR AUC0-inf: number analyzed (Participants) | 15 | 16
  MR AUC0-inf | 4.38 (1.48) | 5.74 (1.79)

31. Secondary Outcome: MR Cmax for N-oxide Voriconazole - Part 3
Description: as for outcome 9
Time Frame: Day 1 of the respective treatment period 1 or 2
Population: as for outcome 2
Measure: Geometric Mean (Standard Deviation); unit: ratio
Arm/Group | Part 3 - ZP-059 | Part 3 - Oral Voriconazole
Number analyzed (Participants) | 16 | 16
ratio | 1.40 (1.44) | 1.84 (1.54)

32. Secondary Outcome: Bioavailability of Voriconazole - Cmax
Description: The Cmax estimated from Part 3 was analyzed to assess the relative bioavailability of inhaled ZP-059 to oral voriconazole.
  The Cmax was compared between asthma subjects in Part 3 and healthy subjects in Part 1 and separately with asthma subjects in Part 2 to assess the relative bioavailability of ZP-059 dose taken in Part 3 in these populations.
  In Part 1 and 3, Cmax was estimated only on Day1. In Part 2, Cmax was estimated on Day 10.
Time Frame: On Day 1 in Parts 1-3 and on Day 10 in Part 2
Population: as for outcome 2
Measure: Geometric Mean (Standard Deviation); unit: ng/mL
Arm/Group | Part 1 - ZP-059 20mg | Part 2 - ZP-059 20mg Bid | Part 3 - ZP-059 | Part 3 - Oral Voriconazole
Number analyzed (Participants) | 6 | 6 | 16 | 16
ng/mL
  Parts 1, 2, and 3 - Day 1 | 53.37 (1.32) | 40.42 (1.33) | 108.08 (1.42) | 863.22 (1.44)
  Part 2 - Day 10: number analyzed (Participants) | 0 | 6 | 0 | 0
  Part 2 - Day 10 |  | 57.11 (1.33) |  |
Statistical Analysis 1: Comparison: Part 3 - ZP-059 vs Part 3 - Oral Voriconazole; Part 3 - ZP-059 20mg: Oral Voriconazole (200mg VFEND); Test type: Other; Geometric mean ratio = 0.13, 90% CI 2-sided [0.107 to 0.146]
Statistical Analysis 2: Comparison: Part 1 - ZP-059 20mg vs Part 3 - ZP-059; ZP-059 20mg: Part 3 / Part 1; Test type: Other; Geometric mean ratio = 2.10, 90% CI 2-sided [1.545 to 2.853]
Statistical Analysis 3: Comparison: Part 2 - ZP-059 20mg Bid vs Part 3 - ZP-059; ZP-059 20mg: Part 3 / Part 2 Day 1; Test type: Other; Geometric mean ratio = 2.63, 90% CI 2-sided [1.953 to 3.544]
Statistical Analysis 4: Comparison: Part 2 - ZP-059 20mg Bid vs Part 3 - ZP-059; ZP-059 20mg: Part 3 / Part 2 Day 10; Test type: Other; Geometric mean ratio = 1.87, 90% CI 2-sided [1.386 to 2.520]

33. Secondary Outcome: Bioavailability of Voriconazole - AUC-inf
Description: The AUC0-inf estimated from Part 3 was analyzed to assess the relative bioavailability of inhaled ZP-059 to oral voriconazole.
  The AUC0-inf was compared between asthma subjects in Part 3 and healthy subjects in Part 1 and separately with asthma subjects in Part 2 to assess the relative bioavailability of ZP-059 dose taken in Part 3 in these populations.
  In Part 1 and 3, AUC0-inf was estimated on Day 1. In part 2, AUC0-in f was estimated on Day 10.
Time Frame: On Day 1 in Parts 1-3 and on Day 10 in Part 2
Population: as for outcome 2
Measure: Geometric Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | Part 1 - ZP-059 20mg | Part 2 - ZP-059 20mg Bid | Part 3 - ZP-059 | Part 3 - Oral Voriconazole
Number analyzed (Participants) | 6 | 6 | 16 | 16
h*ng/mL
  Parts 1, 2, and 3 - Day 1 | 203.96 (1.44) | 155.72 (1.16) | 269.61 (1.56) | 3800.41 (1.92)
  Part 2 - Day 10: number analyzed (Participants) | 0 | 6 | 0 | 0
  Part 2 - Day 10 |  | 258.66 (1.44) |  |
Statistical Analysis 1: Comparison: Part 3 - ZP-059 vs Part 3 - Oral Voriconazole; Part 3 ZP-059 20mg: Oral Voriconazole (200mg VFEND®); Test type: Other; Geometric mean ratio = 0.07, 90% CI 2-sided [0.059 to 0.075]
Statistical Analysis 2: Comparison: Part 1 - ZP-059 20mg vs Part 3 - ZP-059; ZP-059 20mg: Part 3 / Part 1; Test type: Other; Geometric mean ratio = 1.27, 90% CI 2-sided [0.850 to 1.891]
Statistical Analysis 3: Comparison: Part 2 - ZP-059 20mg Bid vs Part 3 - ZP-059; ZP-059 20mg: Part 3 / Part 2 Day 1; Test type: Other; Geometric mean ratio = 2.63, 90% CI 2-sided [1.953 to 3.544]
Statistical Analysis 4: Comparison: Part 2 - ZP-059 20mg Bid vs Part 3 - ZP-059; ZP-059 20mg: Part 3 / Part 2 Day 10; Test type: Other; Geometric mean ratio = 1.87, 90% CI 2-sided [1.386 to 2.520]

ADVERSE EVENTS:
Time Frame: Throughout Part 1 (Day 1, Day 2, Day 3 by phone, Day 5 on return visit) until Days 9-13 by follow-up phone calls. Throughout Part 2 from Day 1 to Day 11, on Day 14 and Day 17 on return visits until Days 11-17 after the last dose by follow-up phone calls. Throughout Part 3 from Day 1 until Day 4
Arm/Group | Part 1 - ZP-059 5mg | Part 1 - ZP-059 10mg | Part 1 - ZP-059 20mg | Part 1 - ZP-059 40mg | Part 2 - ZP-059 10mg Bid | Part 2 - ZP-059 20mg Bid | Part 2 - ZP-059 40mg qd | Part 3 - ZP-059 | Part 3 - Oral Voriconazole
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/16 | 0/16
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/16 | 0/16
Other Adverse Events (participants affected / at risk) | 0/6 | 3/6 | 2/6 | 2/6 | 5/6 | 4/6 | 4/6 | 9/16 | 7/16
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part 1 - ZP-059 5mg (N=6) | Part 1 - ZP-059 10mg (N=6) | Part 1 - ZP-059 20mg (N=6) | Part 1 - ZP-059 40mg (N=6) | Part 2 - ZP-059 10mg Bid (N=6) | Part 2 - ZP-059 20mg Bid (N=6) | Part 2 - ZP-059 40mg qd (N=6) | Part 3 - ZP-059 (N=16) | Part 3 - Oral Voriconazole (N=16)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 2 (2) | 4 (4) | 3 (3)
Migraine (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Stress fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Hot Flush (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dysgeusia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Flatulence (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rhinorrhea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Chest discomfort (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 7 (7) | 1 (1)
Catheter site bruise (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Seasonal allergy (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
FEV decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dysmenorrhoea (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Catheter site pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vessel puncture site pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dizziness postural (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tension headache (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ear discomfort (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2020-06-04): https://cdn.clinicaltrials.gov/large-docs/03/NCT04229303/Prot_000.pdf
  • Statistical Analysis Plan (2020-10-28): https://cdn.clinicaltrials.gov/large-docs/03/NCT04229303/SAP_001.pdf